CLINICAL TRIAL: NCT03954184
Title: Testing of a Patient-centered E-health Implementation Model in Addiction Treatment
Brief Title: E-health Implementation (Iowa)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Iowa (Other); Iowa Department of Public Health (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0997; A195010 (Other: UW-Madison); ENGR/INDUSTRIAL ENGR (Other: UW Madison); 1R01DA044159-01A1 (NIH); 3R01DA044159-02S1 (NIH); Protocol version: 02-15-2021 (Other: Advarra); 2020-0833 (Other: UW Madison (ceded))
Record Dates: First submitted 2019-05-10; First posted 2019-05-17 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU/Control (No Intervention): Sites in the Treatment as Usual (TAU)/Control Arm will receive product training/online support. Sites in the TAU/Control Arm will participate in a one-day product implementation or training session.
- NIATx-TI Framework (Experimental): Sites in the NIATx-TI Arm will receive product training/online support, and training in the NIATx-TI framework. The NIATx-TI framework will include a pre-implementation (planning) phase, and post-implementation (problem-solving) phase, with training delivered by a NIATx-TI coach.
  Interventions: Behavioral: NIATx-TI with Product Training/On-line Support

INTERVENTIONS:
Behavioral: NIATx-TI with Product Training/On-line Support — NIATx-TI framework includes the product training as well as a preimplementation phase and a post-implementation phase. A NIATx-TI coach will provide the training for this arm. The coach will also assist the organizations with applying the NIATx-TI framework.
  Arms: NIATx-TI Framework

SUMMARY:
This research will test a technology adoption framework to increase use of the A-CHESS smartphone app. The project, based in Iowa, will compare a control condition (using a typical product training approach to software implementation that includes user tutorials and instruction on administrative and clinical protocols, followed by access to on-line support) to the typical product training combined with NIATx-TI.

Terms - A-CHESS: Addiction Comprehensive Health Enhancement Support System NIATx-TI: Network for the Improvement of Addiction Treatment-Technology Implementation

DETAILED DESCRIPTION:
Patient-centered e-health has failed to achieve its promise despite considerable consumer interest in technology and research supporting its potential. E-health adoption rates in healthcare are poor, with specialty substance use disorder (SUD) treatment having the lowest technology adoption rate of any sector. Implementation science can address this emerging gap in the e-health field by augmenting existing models, that explain organizational and individual e-health behaviors retrospectively, with prospective models that can guide implementation. The organizational planning discipline, with its decades of research, could provide a cross-disciplinary "jump start" to developing an e-health implementation model for health organizations. Henry Mintzberg, a respected pioneer in this field, describes 2 beneficial approaches to planning: the deliberate approach, which is grounded in pre-implementation planning, and the emergent approach that is grounded in adapting to the environment as the plan is implemented. The proposed e-health implementation model, called the Network for the Improvement of Addiction Treatment-Technology Implementation (NIATx-TI) Framework, incorporates both approaches.

NIATx-TI was piloted in the Iowa Rural Health Information Technology Initiative (IRHIT) with 14 of Iowa's 105 SUD treatment sites and resulted in a 2-fold increase in patients receiving distance treatment. The framework's deliberate component includes using an organizational technology assessment and patient simulation. These tools identify and address assets and barriers to incorporate into the technology's implementation protocol. The framework's emergent component includes using a project team to uncover and prioritize implementation barriers as they arise, develop changes to address identified barriers, and monitor selected adoption measures, while receiving monthly coaching.

This project, based in Iowa, will compare a control condition (using a typical product training approach to software implementation that includes user tutorials and instruction on administrative and clinical protocols, followed by access to on-line support) to the typical product training combined with NIATx-TI. While e-health spans many modalities and health disciplines, this project will focus on the implementing Addiction Comprehensive Health Enhancement Support System (A-CHESS), an evidence-based SUD treatment recovery app developed by our Center for a disease that affects 21.5 million and kills 136,000 Americans annually: substance use disorder. A mobile app was selected, as opposed to another e-health technology, because of the near ubiquitous daily use of mobile technology and because mobile e-health adoption requires supportive participation of both health centers and patients.

In response to the COVID-19 pandemic, the study team added a study component focused on describing how patients are responding to receiving remote treatment (e.g., telehealth). The study team will also seek to understand how using A-CHESS mitigates COVID-19 associated anxiety and loneliness among those with substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18+ years old
* Understand English
* Have a SUD diagnosis
* Have access to a smartphone

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23659 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, Ph.D., Principal Investigator — University of Wisconisn-Madison; David Gustafson, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (49):
- United States (49):
  - Zion Recovery Services, Adel, Iowa
  - Prairie Ridge Integrated Behavioral Healthcare, Algona, Iowa
  - Community and Family Resources, Ames, Iowa
  - Area Substance Abuse Council, Anamosa, Iowa
  - UCS Healthcare, Ankeny, Iowa
  - Zion Recovery Services, Atlantic, Iowa
  - Area Substance Abuse Council, Belle Plaine, Iowa
  - Community and Family Resources, Boone, Iowa
  - Alcohol and Drug Dependency Services (ADDS), Burlington, Iowa
  - Area Substance Abuse Council, Cedar Rapids, Iowa
  - Prairie Ridge Integrated Behavioral Healthcare, Charles City, Iowa
  - Jackson Recovery Centers, Cherokee, Iowa
  - Prelude Behavioral Health Services, Clarence, Iowa
  - Zion Recovery Services, Clarinda, Iowa
  - Community and Family Resources, Clarion, Iowa
  - Heartland Family Services, Council Bluffs, Iowa
  - Area Substance Abuse Council, De Witt, Iowa
  - Jackson Recovery Centers, Denison, Iowa
  - UCS Healthcare, Des Moines, Iowa
  - House of Mercy, Des Moines, Iowa
  - Prelude Behavioral Health Services, Des Moines, Iowa
  - Substance Abuse Services Center, Dubuque, Iowa
  - Prairie Ridge Integrated Behavioral Healthcare, Forest City, Iowa
  - Community and Family Resources, Fort Dodge, Iowa
  - Heartland Family Services, Glenwood, Iowa
  - Zion Recovery Services, Greenfield, Iowa
  - Prairie Ridge Integrated Behavioral Healthcare, Hampton, Iowa
  - Community and Family Resources, Humboldt, Iowa
  - House of Mercy, Indianola, Iowa
  - Prelude Behavioral Services, Iowa City, Iowa
  - ADDS, Keokuk, Iowa
  - UCS Healthcare, Knoxville, Iowa
  - Jackson Recovery Centers, Le Mars, Iowa
  - Heartland Family Services, Logan, Iowa
  - Area Substance Abuse Council, Maquoketa, Iowa
  - Prelude Behavioral Health Services, Marengo, Iowa
  - Prairie Ridge Integrated Behavioral Healthcare, Mason City, Iowa
  - ADDS, Mount Pleasant, Iowa
  - House of Mercy, Newton, Iowa
  - Zion Recovery Services, Perry, Iowa
  - Community and Family Resources, Pocahontas, Iowa
  - Zion Recovery Services, Red Oak, Iowa
  - Community and Family Resources, Rockwell City, Iowa
  - Zion Recovery Services, Shenandoah, Iowa
  - Jackson Recovery Centers, Sioux City, Iowa
  - Prelude Behavioral Services, Tipton, Iowa
  - Area Substance ABuse Council, Vinton, Iowa
  - ADDS, Wapello, Iowa
  - Community and Family Resources, Webster City, Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fleddermann K, Molfenter T, Vjorn O, Horst J, Hulsey J, Kelly B, Zawislak K, Gustafson DH, Gicquelais RE. Patient Preferences for Mobile Health Applications to Support Recovery. J Addict Med. 2023 Jul-Aug 01;17(4):394-400. doi: 10.1097/ADM.0000000000001137. Epub 2023 Jan 18. PMID 37579096
- [Result] Fleddermann K, Molfenter T, Jacobson N, Horst J, Roosa MR, Boss D, Ross JC, Preuss E, Gustafson DH. Clinician Perspectives on Barriers and Facilitators to Implementing e-Health Technology in Substance Use Disorder (SUD) Treatment Facilities. Subst Abuse. 2021 Oct 26;15:11782218211053360. doi: 10.1177/11782218211053360. eCollection 2021. PMID 34720585
- [Derived] Gustafson D Sr, Horst J, Boss D, Fleddermann K, Jacobson N, Roosa M, Ross JC, Gicquelais R, Vjorn O, Siegler T, Molfenter T. Implementation of Smartphone Systems to Improve Quality of Life for People With Substance Use Disorder: Interim Report on a Randomized Controlled Trial. JMIR Hum Factors. 2022 Jul 14;9(3):e35125. doi: 10.2196/35125. PMID 35834315
- [Derived] White VM, Molfenter T, Gustafson DH, Horst J, Greller R, Gustafson DH Jr, Kim JS, Preuss E, Cody O, Pisitthakarm P, Toy A. NIATx-TI versus typical product training on e-health technology implementation: a clustered randomized controlled trial study protocol. Implement Sci. 2020 Oct 23;15(1):94. doi: 10.1186/s13012-020-01053-4. PMID 33097097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (SUD clinic sites) funded by the Iowa Department of Health and Human Services (formerly Iowa Department of Public Health) were recruited between May 2019 and April 2020.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | TAU/Control | NIATx-TI Framework
Started | 11086; 20 Clinics | 12573; 21 Clinics
Patients | 10972; 20 Clinics | 12379; 21 Clinics
Counselors | 114; 20 Clinics | 194; 21 Clinics
Completed | 10586; 19 Clinics (10472 patient participants completed, 114 counselors completed.) | 12573; 21 Clinics (12379 patient participants and 194 counselor participants completed.)
Not Completed | 500; 1 Clinics | 0; 0 Clinics
Not completed — Lost to Follow-up | 500 | 0

BASELINE CHARACTERISTICS:
Population: For each of our sites (19 control and 21 intervention) we have population data collected from Iowa department of public health and each site.
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | TAU/Control | NIATx-TI Framework | Total
Number analyzed (Participants) | 10586 | 12573 | 23159
Number analyzed (Clinics) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was collected from the Iowa department of public health as well as the sites. Population: Patient participants and counselors were counted separately.
  years
    Participants: number analyzed (Participants) | 10472 | 12379 | 22851
    Participants | 34.8 (12.2) | 36.0 (12.4) | 35.5 (12.3)
    Counselors: number analyzed (Participants) | 114 | 194 | 308
    Counselors | 42.4 (11.5) | 45.1 (12.4) | 44.3 (12.2)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender was collected for patients from the Iowa department of public health. For counselors this data was gathered from the sites. Population: Gender was collected for patients and counselors separately.
  Participants
    Patients: Genderqueer/Other: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Genderqueer/Other | 5 | 73 | 78
    Patients: Man: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Man | 5192 | 7623 | 12815
    Patients: Refused/Unknown: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Refused/Unknown | 2564 | 445 | 3009
    Patients: Transgender Man: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Transgender Man | 5 | 3 | 8
    Patients: Transgender Woman: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Transgender Woman | 3 | 6 | 9
    Patients: Woman: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Woman | 2703 | 4229 | 6932
    Counselors: Genderqueer/Other: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Genderqueer/Other | 0 | 0 | 0
    Counselors: Man: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Man | 10 | 48 | 58
    Counselors: Refused/Unknown: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Refused/Unknown | 3 | 30 | 33
    Counselors: Transgender Man: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Transgender Man | 0 | 0 | 0
    Counselors: Transgender Woman: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Transgender Woman | 0 | 0 | 0
    Counselors: Woman: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Woman | 101 | 116 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was collected for patients from the Iowa department of public health. For counselors this data was gathered from the sites. Population: Patients and counselors were analyzed separately. The numbers analyzed in each arm for each row do add up to the overall number analyzed.
  Participants
    Patients: number analyzed (Participants) | 10472 | 12379 | 22851
    Patients: Hispanic or Latino | 926 | 674 | 1600
    Patients: Not Hispanic or Latino | 8920 | 11212 | 20132
    Patients: Unknown or Not Reported | 626 | 493 | 1119
    Counselors: number analyzed (Participants) | 114 | 194 | 308
    Counselors: Hispanic or Latino | 2 | 6 | 8
    Counselors: Not Hispanic or Latino | 98 | 118 | 216
    Counselors: Unknown or Not Reported | 14 | 70 | 84
Region of Enrollment [Number; unit: participants]
  United States | 10586 | 12573 | 23159
Average # of admissions [Mean (Standard Deviation); unit: Number of admissions] | 68.2 (82.6) | 78.3 (111.6) | 73.5 (97.8)
Site location (rural v urban) [Number; unit: Number of sites]
  Rural | 1 | 3 | 4
  Urban | 17 | 17 | 34
  Half Rural/ Half Urban | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Reach: As Assessed by the Mean Number of Clinics With Participants Who Download the A-CHESS App
Description: The mean number of clinics with patients who download the A-CHESS app will be obtained monthly during the study via the A-CHESS server and Iowa Department of Public Health (IDPH) data.
Time Frame: 45 months
Measure: Mean (Standard Error); unit: Mean number of clinics
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 19 | 21
Mean number of clinics | 0.039 (0.029) | 0.171 (0.041)

2. Primary Outcome: Reach: As Assessed by the Number of Days That Participants Use the A-CHESS
Description: The frequency of use of A-CHESS by each participant will be obtained monthly during the study via the A-CHESS server and Iowa Department of Public Health (IDPH) data.
Time Frame: 45 months
Population: 6 sites are excluded from the analysis because they are comprised entirely of patients without activated accounts.
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 14 | 20
Days | 0.161 (0.466) | 1.845 (1.487)

3. Secondary Outcome: Effectiveness of A-CHESS as Assessed by the Retention Rate of Eligible Participants.
Description: Retention rates of eligible participants
Time Frame: Collected monthly during months 13 - 45
Population: This data was not collected
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adoption: Number of Days Each Counselor Used the A-CHESS
Description: Number of days each counselor used the A-CHESS will be assessed by A-CHESS logs
Time Frame: 45 months
Population: Those counselors that did not use RISE at least once were not included in this calculation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 89 | 100
days | 1.81 (2.52) | 19.11 (62.68)

5. Secondary Outcome: Adoption - The Percentage of Counselors Using A-CHESS Will be Assessed Via the Organizational Survey and A-CHESS Logs
Description: Organizational survey will be completed by a member of the management team two times during the project (organizational baseline, end of the intervention)
Time Frame: Collected twice during study; starting M22 - 31 and M35-44
Population: Any counselor who had the opportunity to have patients connected to them in the app is counted in the overall number
Measure: Count of Participants; unit: Participants
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 110 | 193
Participants | 24 | 84

6. Secondary Outcome: A-CHESS/NIATx Implementation Fidelity (Survey)
Description: Survey data on participating organizations' fidelity to the NIATx Technology Implementation (NIATx-TI) process. The Implementation Fidelity survey is a 13 item questionnaire using a 4-point scale where 0 = Not True and 4 = True. Scores range from 0-52. Higher scores indicate greater implementation fidelity.
Time Frame: Collected twice during study; approx. M14 - 25 and M32 - 43
Population: Not all sites completed surveys at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 17 | 20
score on a scale
  Survey 2 | 2.26 (0.55) | 2.91 (0.51)
  Survey 3 | 2.20 (0.63) | 2.91 (0.55)

7. Secondary Outcome: Organizational Readiness of Participating Organizations as Assessed by Organizational Change Manager (Survey)
Description: Survey data on the organizational readiness of participating organizations. Organizational Readiness (as measured by Organizational Change Manager) - 5 categories from Not True (0) to True (3) and Don't Know (No score). Scores range from 0-66. Higher scores indicate greater readiness for change.
Time Frame: Collected twice during study; approx. M14 - 25 and M32 - 43
Population: Not all sites completed all surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 17 | 20
score on a scale
  Survey 2 | 2.99 (0.58) | 3.17 (0.50)
  Survey 3 | 2.73 (0.75) | 3.28 (0.40)

8. Secondary Outcome: Financial Resource Availability (Survey)
Description: Survey data on how the organization's financial resource availability affects A-CHESS implementation. Scored the availability of financial resources on a 5-point scale from 0= Not Ture to 4= True. Scores range from 0-28. Higher score indicates greater availability of resources.
Time Frame: Collected twice during study; starting M22 - 31 and M35-44
Population: Not all sites completed all surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 17 | 21
units on a scale
  Survey 1 | 2.68 (0.73) | 3.41 (0.57)
  Survey 2 | 2.77 (0.83) | 3.13 (0.87)

9. Secondary Outcome: Difference in Number of Admissions in Rural vs. Urban Location
Description: Statistical analysis of organizational traits will be done by calculating the difference in number of admissions in rural vs. urban location. The number of clinics located in a rural area was counted. The number of clinics in an urban location were counted.
Time Frame: Collected during months 7, 18, 30, and 42, month 42 reported
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | TAU/Control | NIATx-TI Framework
Number analyzed (Participants) | 10586 | 12573
Number analyzed (Clinics) | 19 | 21
Clinics
  Rural | 1 | 3
  Urban | 17 | 17
  Half Rural/ Half Urban | 1 | 1

10. Other Pre Specified Outcome: Supplement 1 - Understand Impact of ACHESS on pt Anxiety and Loneliness During COVID-19 Pandemic
Description: Online survey
Time Frame: M34-37
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Supplement 2 - Understand How Treatment Organizations and Staff Used ACHESS During COVID Pandemic
Description: Online survey
Time Frame: M34-37
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months (1 year, 6 months)
Arm/Group | TAU/Control | NIATx-TI Framework
All-Cause Mortality (participants affected / at risk) | 0/10586 | 0/12573
Serious Adverse Events (participants affected / at risk) | 0/10586 | 0/12573
Other Adverse Events (participants affected / at risk) | 0/10586 | 0/12573

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT03954184/Prot_SAP_000.pdf